CLINICAL TRIAL: NCT06401265
Title: Recalling the Treatment and Prognosis of Upper Tract Urothelial Cancer (UTUC)
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 06-X34-105
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2022-02

CONDITIONS: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among urothelial cancers, upper urinary tract urothelial cancers, including renal pelvis and ureteral cancers have a higher incidence rate in Taiwan than Western countries. In particular, the proportion of female patients is similar to that of males. This situation is significantly different from that in foreign countries. The cause is currently uncertain.In the past, the arsenic contamination of groundwater made blackfoot disease become common and malignant in areas. Now, the number of kidney dialysis patients in Taiwan is increasing; and according to statistics, there is a significantly higher incidence of urothelial cancer among kidney dialysis patients. This may be caused by the use of traditional Chinese medicine or other unknown reasons.

ELIGIBILITY:
Inclusion Criteria:

* Case study of upper urinary tract urothelial cancer surgery

Exclusion Criteria:

* Cases of surgery for non-upper urinary tract urothelial cancer

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with upper urinary tract urothelial carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
It is a retrospective and questionnaire-based study. | Patients with urothelial carcinoma of the upper urinary tract from January 2008 to December 2019.

CONTACTS AND LOCATIONS:
Locations (1):
- Tzu Chi hospital, Taipei, Taiwan